CLINICAL TRIAL: NCT04532333
Title: Anticoagulant Efficacy and Safety of BivalirUdin Versus heparIn During coiL Embolization in Patients With ruptureD Intracranial Aneurysms: an Open-label, Multicenter, Randomized Pilot Study（BUILD）
Brief Title: Efficacy and Safety of Bivalirudin Versus Heparin During Coil Embolization in Patients With Ruptured Intracranial Aneurysms
Acronym: BUILD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Zhejiang University (Other); Wuhan University (Other); Qilu Hospital of Shandong University (Other); The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Dean of Neurosurgical Department,Changhai Hospital,Shanghai,China, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHEC2020-042
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Anticoagulant Agents; Aneurysm, Intracranial Berry; Therapeutic Embolization; Anticoagulation Agents; Heparin Sodium; Bivalirudin
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm | interventions — bivalirudin; Injections; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin at full dose Bivalirudin 0.75 mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until end of the procedure
  Interventions: Drug: Bivalirudin 250 MG Injection
- Heparin (Active Comparator): Heparin first dose at 0.6mg/kg(75U/kg) Heparin should be administered each hour, 0.6mg/kg(75U/kg) as bolus dose, 0.3mg/kg 1h later, 10mg(1250U) every hour after.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin 250 MG Injection — Bivalirudin 0.75 mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until end of the procedure
  Arms: Bivalirudin
Drug: Heparin — Heparin should be administered each hour, 0.6mg/kg(75U/kg) as bolus dose, 0.3mg/kg 1h later, 10mg(1250U) every hour after.
  Arms: Heparin

SUMMARY:
This is a randomized, open label, multi-center, positive-controlled study, in which a total of 236 patients will be enrolled and randomly assigned to receive bivalirudin or heparin in a 1:1 ratio during coil embolization in patients with ruptured intracranial aneurysms.

Procedure-related complication, mRS, Activated Clotting Time, ischemic and hemorrhagic complications, symptomatic and asymptomatic intracranial hemorrhage, death, Heparin Induced Thrombocytopenia will be evaluated during procedure, at 24hs, 7days and 30 days after.

DETAILED DESCRIPTION:
Endovascular embolization has become an effective modality for the treatment of intracranial aneurysms. Despite advances in technology and techniques, thromboembolic and bleeding events are still encountered as inherent perioperative complications. Hypercoagulability as a systemic response to acute subarachnoid hemorrhage (SAH) may be associated with an increased incidence of thromboembolic events.

The administration of anticoagulant may reduce thromboembolic events during the endovascular embolization, meanwhile, involves the risk of bleeding. Although heparin is commonly used during the procedure, the safety in patients with ruptured intracranial aneurysms has not been established. In contrast to heparin, bivalirudin is a short-lived direct thrombin inhibitor with an intrinsic antiplatelet activity and more stable pharmacokinetic and pharmacodynamic properties which has been associated with reduced bleeding and an overall favorable profile. Bivalirudin administration in patients with high bleeding risk during coronary intervention is recommended by current guidelines.

This is an open label, multicenter, randomized pilot study, which is aimed to investigate the safety and efficacy of bivalirudin coil embolization in patients with ruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years, any gender
* intracranial aneurysms ruptured in 14 days
* Diagnosed as subarachnoid hemorrhage (SAH) by CT, confirmed aneurysmal SAH by DSA
* Hunt-Hess I-III
* Patient is suitable for coil embolization
* Informed consent and availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements

Exclusion Criteria:

* Nonsaccular Aneurysms (include infective, fusiform, dissecting aneurysms)
* Prior intracranial aneurysms
* Poor baseline of mRS 4-5
* Aneurysms that cannot be successfully treated by interventional treatment judged by clinician.
* Patients cannot receive antiplatelet aggregation or anticoagulant therapy
* Patients with indications for emergency craniotomy: intracranial hematoma, high intracranial pressure or hydrocephalus etc..
* Patients with AVM, intracranial artery stenosis or moyamoya disease
* Pregnancy or lactation
* Patients with severe abnormal function of main organs, liver or kidney
* Other serious diseases not suitable for this study
* Patients are currently participating in another drug-related clinical study
* Patients are allergic to heparin or bivalirudin and its excipients or hirudin
* Patients with a clear history of allergy to coil embolic material
* Patients had or may have had severe reactions to contrast media that could not complete the preoperative medication
* Patients are not suitable to participate in this clinical study judged by clinician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Procedure-related complication | 30 days
  A composite of of death from any cause, thromboembolic events, or bleeding defined by BARC definition 3 or 5 BARC=Bleeding Academic Research Consortium

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 30 days
  The mRS score, and proportion of subjects achieving mRS score of 0-2
Activated Clotting Time (ACT) | During procedure
  ACT values of 0 min and 5 min after bolus injection will be recorded in all patients Extra ACT values of 15 min, 30 min, 55min, 65 min,and 115 min after bolus injection will be recorded in 8 patients of both arm, and the curve will be simulated
Procedure-related complication | During procedure, at 24hs, 7days
  A composite of of death from any cause, thromboembolic events, or bleeding defined by BARC definition 3 or 5 BARC=Bleeding Academic Research Consortium
Thromboembolic events | During procedure, at 24hs, 7days, 30days
  Definition:
  1. Intraoperative: stent thrombosis/stenosis, distal vascular occlusion on imaging
  2. Postoperative： 1) new deficits or change in level of consciousness, intracranial hemorrhage cause is excluded by CT, 2) no clinical symptom but CT showed new infarction
Bleeding events | During procedure, at 24hs, 7days, 30days
  Any bleeding as defined by the BARC definition (except grade 4) Any bleeding as defined by the GUSTO definition
Intracranial hemorrhage | During procedure, at 24hs, 7days, 30days
  Intracranial hemorrhage and Symptomatic intracranial hemorrhage
Heparin-induced thrombocytopenia(HIT) | 7days
  defined as a platelet count decrease ofmore than50%or more than 150 × 109/L frombaseline

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, M.D., Principal Investigator — Neurosurgical Department of Changhai Hospital; Sheng Guan, M.D., Principal Investigator — Neurointerventional Department, The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: Undecided